CLINICAL TRIAL: NCT00922844
Title: The Effect of Sevoflurane Versus Isoflurane on Vasopressor Need
Acronym: ESIVAN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: too slow recruitment; lack of funding
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, D van Dijk, Dr, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL24375.041.08
Record Dates: First submitted 2009-06-12; First posted 2009-06-17 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Hypotension
Keywords: hypotension; low blood pressure; vasopressor need
MeSH Terms: conditions — Hypotension | interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Active Comparator): Administration of the volatile anesthetic Sevoflurane.
  Interventions: Drug: Sevoflurane and isoflurane
- Isoflurane (Active Comparator): Administration of the volatile anesthetic Isoflurane.
  Interventions: Drug: Sevoflurane and isoflurane

INTERVENTIONS:
Drug: Sevoflurane and isoflurane — Patients will be randomized to a 10 minute treatment with isoflurane, followed by a wash-out period, followed by a 10 minute treatment with sevoflurane, or the other way round.
  Other Names: Sevorane/isoflurane

SUMMARY:
Aim of this study is to determine the effect of isoflurane versus sevoflurane on blood pressure and systemic vascular resistance.

DETAILED DESCRIPTION:
In modern anesthesia a variety of volatile anesthetics is available. In cardiac anesthesiology both isoflurane and sevoflurane are frequently used. At present the number of studies comparing the influence of isoflurane and sevoflurane on blood pressure and systemic vascular resistance is limited. Moreover, the results presented in the available literature are inconsistent. The decision as to which of both volatiles should be used during cardiac surgery is not evidence-based, but is based on personal preference of the anesthesist. The most reliable way to compare the effects of isoflurane and sevoflurane on blood pressure and systemic vascular resistance is a randomized controlled trial in patients during Cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* competent adult patients (18 years or older)undergoing elective coronary artery bypass grafting with the use of the cardiopulmonary bypass.

Exclusion Criteria:

* Patients undergoing valve surgery or combined surgical procedures (e.g. coronary artery bypass grafting in combination with valve reconstruction.
* uncontrolled hypertension
* a poor left ventricular function
* renal failure
* a body mass index of > 25
* history of cerebrovascular accident, transient ischemic accident or carotid artery stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Total amount of the vasopressor phenylephrine that is needed to maintain blood pressure above 60 mmHg during 10 minutes of Cardiopulmonary bypass. | 10 minutes

SECONDARY OUTCOMES:
Mean blood pressure throughout the 10 minute periods, the need for a stronger vasopressor (norepinephrine) and the inability to keep mean blood pressure below 75 mmHg at MAC 0.6. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: C.J. Kalkman, MD, PhD, Study Chair — UMC Utrecht
Locations (1):
- University Medical Center, Utrecht, Utrecht, Netherlands